CLINICAL TRIAL: NCT02167893
Title: Leuprorelin Acetate SR 11.25 mg Injection Kit Specified Drug-use Survey "Long-term Use Survey in Prostate Cancer Patients (96 Weeks)"
Brief Title: Leuplin SR 11.25 mg Injection Kit Specified Drug-use Survey "Long-term Use Survey in Prostate Cancer Patients (96 Weeks)"
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: 265-021; JapicCTI-142560 (Registry Identifier: JapicCTI); JapicCTI-R160837 (Other: JapicCTI)
Record Dates: First submitted 2014-06-17; First posted 2014-06-19 (Estimated); Results first posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-02

CONDITIONS: Prostate Cancer
Keywords: Pharmacological therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Leuprolide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subcutaneous administration of leuprorelin acetate: Subcutaneous administration of leuprorelin acetate once every 12 weeks as daily medicinal practice.
  Interventions: Drug: Leuprorelin acetate

INTERVENTIONS:
Drug: Leuprorelin acetate — Leuprorelin acetate SR 11.25 mg injection kit
  Other Names: Leuplin SR 11.25 mg Injection Kit

SUMMARY:
The purpose of this survey is designed to evaluate the efficacy and safety of long-term use (96 weeks) of leuprorelin acetate SR 11.25 milligram (mg) injection kit (Leuplin SR 11.25 mg injection kit) in prostate cancer participants in daily medical practice.

DETAILED DESCRIPTION:
This survey was designed to evaluate the efficacy and safety of long-term use (96 weeks) of leuprorelin acetate 3 months depot injection kit (Leuplin SR 11.25 mg Injection Kit) in prostate cancer participants in daily medical practice.

For adults, 11.25 mg of leuprorelin acetate is usually administered subcutaneously once every 12 weeks. Prior to injection, the plunger rod of the syringe is pushed upward with the needle pointed upward, allowing the entire suspension fluid contained to be transferred to the powder. The powder is then fully suspended in the fluid while ensuring that bubbles are not generated.

ELIGIBILITY:
Inclusion Criteria: Prostate cancer participants who meet all the following criteria:

1. Participants for whom prostate cancer was initially diagnosed on or after January 1, 2005
2. Participants with no prior history of treatment with Leuplin SR 11.25 mg Injection Kit (as an exception, participants with prior history of treatment with Leuplin 3.75 mg Injection Kit may be enrolled in the survey )
3. Participants with prostate-specific antigen (PSA) level determined at baseline or within 3 months prior to the start of treatment with Leuplin SR 11.25 mg Injection Kit

Exclusion Criteria:

-

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 11288 (Actual)
Dates: Start 2005-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Postmarketing Group Manager, Study Chair — Takeda

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 758 investigative site in Japan from 13-Oct-2005 to 31-Dec-10.
Pre-assignment Details: Participants with a historical diagnosis of prostate cancer were treated with leuprorelin acetate 11.25 milligrams (mg) in daily medical practice along with adjuvant therapy were observed.
Groups:
- Leuprorelin Acetate: Participants receiving leuprorelin acetate 11.25 mg, injection subcutaneously once every 12 weeks up to 96 weeks as daily medical practice were observed.
Period: Overall Study
Arm/Group | Leuprorelin Acetate
Started | 11288
Completed | 11125
Not Completed | 163
Not completed — Investigator transferred | 85
Not completed — Investigator health reasons | 10
Not completed — Case report forms not collected | 68

BASELINE CHARACTERISTICS:
Population: The safety analysis set was defined as all participants who were enrolled and completed the study.
Arm/Group | Leuprorelin Acetate
Number analyzed (Participants) | 11125
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.88 (7.04)
Sex/Gender, Customized [Number; unit: participants]
  Male | 11125
Body Mass Index [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 22.87 (3.10)
Tumor Node Metastasis(TNM) Classification (at start of treatment with leuplin SR 11.25 mg injection) [Number; unit: participants] — TNM classification based on tumor size, if cancer cells had spread to nearby lymph nodes (LN), or distant metastasis. Stages included: stage 0(no evidence of cancer cells),stage 1(T1N0M0), stage IIA(T0N1M0, T1N1M0, T2N0M0), stage IIB(T2N1M0, T3N0M0), stage IIIA(T0N2M0, T1N2M0, T2N3M0, T3N1orN2M0),stage IIIb( T4 anyNM0, any TN3M0),stage IIIC(any TN3M0), stage IV(any T any NM1), where T0=early form of tumor, T1=<2 centimeter (cm), T2=2-5 cm, T3=>2 cm, T4=large sized, N0=not spread to LN, N1=spread to 1 to 3,N2=spread to 4 to 9,N3=spread >10 axillary LN, M0=no metastasis, M1= Metastasis.
  participants
    No lesions | 333
    Stage I | 529
    Stage II | 5197
    Stage III | 2066
    Stage IV | 2608
    Cannot be assessed | 391
    Unknown | 1
Performance Status (at start of treatment with leuplin SR 11.25 mg injection) [Number; unit: participants] — Following are ECOG grades. 0: Fully active, perform all pre-disease activities without restriction. 1: Restricted in physically strenuous activity but ambulatory, carry out work of a light or sedentary nature. 2: Ambulatory, capable of selfcare, unable to carry out any work activities, up and about more than (>) 50% of waking hours. 3: Capable of limited selfcare, confined to bed or chair >50% of waking hours. 4: Completely disabled, not capable of any selfcare, totally confined to bed or chair.
  participants
    0 | 8577
    1 | 1688
    2 | 518
    3 | 230
    4 | 72
    Unknown | 40
Predisposition to Hypersensitivity [Number; unit: participants]
  Had predisposition to Hypersensitivity | 530
  Had no redisposition to Hypersensitivity | 10594
  Unknown | 1
Medical Complications [Number; unit: participants] — Participants may be represented in more than 1 category.
  participants
    Had Complications | 7234
    Had no Complications | 3889
    Unknown | 2
Breakdown of Complications [Number; unit: participants] — This baseline characteristic was analyzed in participants who had hypertension, heart disease, diabetes mellitus, hyperlipidemia, malignant tumor, cerebrovascular disease, and any other medical complications.
  participants
    Hypertension | 3195
    Heart disease | 1208
    Diabetes mellitus | 1147
    Hyperlipidemia | 799
    Cerebrovascular disease | 547
    Malignant tumor | 456
    Other | 4617
Prior Treatment for Prostate Cancer [Number; unit: participants] — This baseline measure was analyzed in participants who had treatment for prostate cancer prior to the start of treatment with leuplin SR 11.25 mg. Participants may be represented in more than 1 category.
  participants
    Had prior treatment | 9324
    Had no prior treatment | 1799
    Unknown | 2
Breakdown for Prior Treatment for Prostate Cancer [Number; unit: participants] — LH-RH (luteinizing hormone releasing hormone)
  participants
    LH-RH agonists (other than leuplin SR 11.25 mg) | 7220
    Other endocrine therapies | 7596
    Other chemotherapies | 49
    Total prostatectomy | 734
    Radiotherapy | 561
    Other treatments | 72
Healthcare Category [Number; unit: participants] — Participants were categorized as outpatient and inpatient.
  participants
    Outpatient | 10629
    Inpatient | 496

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting One or More Adverse Drug Reactions
Description: Adverse drug reactions are defined as adverse events (AEs) which are in the investigator's opinion of causal relationship to the study treatment. AEs are defined as any unfavorable and unintended signs, symptoms or diseases temporally associated with the use of a medicinal product reported from the first dose of study drug to the last dose of study drug.
Time Frame: Baseline up to Week 96
Population: The safety analysis set was defined as all participants who were enrolled and completed the study.
Measure: Number; unit: participants
Arm/Group | Leuprorelin Acetate
Number analyzed (Participants) | 11125
participants | 2052

2. Primary Outcome: Number of Participants Reporting One or More Serious Adverse Drug Reactions
Description: Serious adverse drug reactions are defined as serious adverse events (SAE) which are in the investigator's opinion of causal relationship to the study treatment. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Baseline up to Week 96
Population: The safety analysis set was defined as all participants who were enrolled and completed the study.
Measure: Number; unit: participants
Arm/Group | Leuprorelin Acetate
Number analyzed (Participants) | 11125
participants | 188

3. Secondary Outcome: Percentage of Participants With Progression Free Survival (PFS) Based on TNM Classification
Description: PFS was defined as the time from the first day of study treatment to documented disease progression or death on study. For participants who experienced no disease progression and did not die while on study, data were censored at the date of the last tumor assessment. Kaplan-Meier methodology was used to estimate PFS. TNM classification based on tumor size, if cancer cells had spread to nearby lymph nodes (LN), or distant metastasis. Stages included: stage 0(no evidence of cancer cells),stage 1(T1N0M0), stage IIA(T0N1M0, T1N1M0, T2N0M0), stage IIB(T2N1M0, T3N0M0), stage IIIA(T0N2M0, T1N2M0, T2N3M0, T3N1orN2M0),stage IIIb( T4 anyNM0, any TN3M0),stage IIIC(any TN3M0), stage IV(any T any NM1), where T0=early form of tumor, T1=<2 centimeter (cm), T2=2-5 cm, T3=>2 cm, T4=large sized, N0=not spread to LN, N1=spread to 1 to 3,N2=spread to 4 to 9,N3=spread >10 axillary LN, M0=no metastasis, M1= Metastasis.
Time Frame: Baseline up to 96 weeks
Population: The efficacy assessment population was defined as all participants whose efficacy data at baseline and at least 1 post-baseline time points was available.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Leuprorelin Acetate
Number analyzed (Participants) | 9691
percentage of participants
  Stage I (N=467) | 94.2 [91.4 to 96.2]
  Stage II (N=4852) | 92.0 [91.2 to 92.8]
  Stage III (N=1926) | 86.9 [85.2 to 88.4]
  Stage IV (N=2446) | 55.4 [53.3 to 57.5]

4. Secondary Outcome: Percentage of Participants With Overall Survival (OS) Based on TNM Classification
Description: OS was defined as the duration from randomization to death (due to any cause). Probability of OS was reported using Kaplan-Meier method. TNM classification based on tumor size, if cancer cells had spread to nearby lymph nodes (LN), or distant metastasis. Stages included: stage 0(no evidence of cancer cells),stage 1(T1N0M0), stage IIA(T0N1M0, T1N1M0, T2N0M0), stage IIB(T2N1M0, T3N0M0), stage IIIA(T0N2M0, T1N2M0, T2N3M0, T3N1orN2M0),stage IIIb( T4 anyNM0, any TN3M0),stage IIIC(any TN3M0), stage IV(any T any NM1), where T0=early form of tumor, T1=<2 centimeter (cm), T2=2-5 cm, T3=>2 cm, T4=large sized, N0=not spread to LN, N1=spread to 1 to 3,N2=spread to 4 to 9,N3=spread >10 axillary LN, M0=no metastasis, M1= Metastasis.
Time Frame: Baseline up to 96 weeks or death (which ever occurs first)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Leuprorelin Acetate
Number analyzed (Participants) | 9688
percentage of participants
  Stage I (N=466) | 96.9 [94.6 to 98.2]
  Stage II (N=4852) | 97.4 [96.8 to 97.8]
  Stage III (N=1927) | 97.6 [96.7 to 98.2]
  Stage IV (N=2443) | 88.5 [87.0 to 89.8]

5. Secondary Outcome: Percentage of Participants With Metastasis-free Survival
Time Frame: Baseline up to 96 weeks
Population: No results have been reported in this measure because as predefined in the protocol, the outcome measure was not planned to be assessed.
Arm/Group | Leuprorelin Acetate
Number analyzed (Participants) | 0

6. Secondary Outcome: Percentage of Participants With Disease-specific Survival
Description: Disease-specific survival is defined as time interval between the date of randomization and the earliest date of local, regional or distant relapse, or death due to cancer.
Time Frame: Baseline up to 96 weeks
Population: as for outcome 5
Arm/Group | Leuprorelin Acetate
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 96 weeks
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Only adverse drug reactions were collected in this study.
Arm/Group | Leuprorelin Acetate
Serious Adverse Events (participants affected / at risk) | 188/11125
Other Adverse Events (participants affected / at risk) | 1429/11125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Leuprorelin Acetate (N=11125)
Gastroenteritis (Infections and infestations) | 2
Herpes zoster (Infections and infestations) | 1
Injection site abscess (Infections and infestations) | 6
Lung abscess (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 10
Pyelonephritis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Pseudomonas infection (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Marasmus (Metabolism and nutrition disorders) | 2
Decreased appetite (Metabolism and nutrition disorders) | 4
Hyperlipidaemia (Metabolism and nutrition disorders) | 1
Delirium (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Altered state of consciousness (Nervous system disorders) | 3
Cerebellar haemorrhage (Nervous system disorders) | 1
Cerebellar infarction (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 16
Cerebrovascular disorder (Nervous system disorders) | 1
Dementia (Nervous system disorders) | 4
Dysarthria (Nervous system disorders) | 2
Dyslalia (Nervous system disorders) | 2
Embolic stroke (Nervous system disorders) | 2
Hemiplegia (Nervous system disorders) | 2
Hyperreflexia (Nervous system disorders) | 1
Optic neuritis (Nervous system disorders) | 1
Speech disorder (Nervous system disorders) | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Facial nerve disorder (Nervous system disorders) | 1
Thrombotic cerebral infarction (Nervous system disorders) | 1
Cataract (Eye disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 9
Cardiac failure acute (Cardiac disorders) | 2
Cardio-respiratory arrest (Cardiac disorders) | 2
Cardiomegaly (Cardiac disorders) | 3
Myocardial infarction (Cardiac disorders) | 4
Cardiac failure congestive (Cardiac disorders) | 3
Myocardial ischaemia (Cardiac disorders) | 1
Prinzmetal angina (Cardiac disorders) | 1
Ventricular hypokinesia (Cardiac disorders) | 1
Cardiac disorder (Cardiac disorders) | 1
Aortic aneurysm (Vascular disorders) | 2
Hypertension (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Hot flush (Vascular disorders) | 1
Arteriosclerosis obliterans (Vascular disorders) | 1
Aortic dissection rupture (Vascular disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 9
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 1
Nocturnal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Abdominal pain lower (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diverticulum intestinal (Gastrointestinal disorders) | 1
Faeces discoloured (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 2
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 2
Melaena (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Gallbladder perforation (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 5
Liver disorder (Hepatobiliary disorders) | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Generalised erythema (Skin and subcutaneous tissue disorders) | 1
Incontinence (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Asthenia (General disorders) | 1
Chest discomfort (General disorders) | 1
Chest pain (General disorders) | 1
Crepitations (General disorders) | 3
Death (General disorders) | 13
Face oedema (General disorders) | 1
Gait disturbance (General disorders) | 3
Injection site erosion (General disorders) | 1
Injection site erythema (General disorders) | 12
Injection site haemorrhage (General disorders) | 1
Injection site induration (General disorders) | 11
Injection site pain (General disorders) | 9
Injection site pruritus (General disorders) | 4
Injection site ulcer (General disorders) | 3
Injection site warmth (General disorders) | 1
Malaise (General disorders) | 1
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 4
Injection site swelling (General disorders) | 10
Alanine aminotransferase increased (Investigations) | 6
Aspartate aminotransferase increased (Investigations) | 6
Blood cholesterol increased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Blood triglycerides increased (Investigations) | 1
C-reactive protein increased (Investigations) | 1
Chest X-ray abnormal (Investigations) | 3
Computerised tomogram abnormal (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Haemoglobin decreased (Investigations) | 2
Low density lipoprotein increased (Investigations) | 1
Platelet count decreased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Surfactant protein increased (Investigations) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Compression fracture (Injury, poisoning and procedural complications) | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 3
Forearm fracture (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 4
Cardiac pacemaker insertion (Surgical and medical procedures) | 1
Hospitalisation (Surgical and medical procedures) | 2
Acute myocardial infarction (Cardiac disorders) | 3
Angina pectoris (Cardiac disorders) | 5
Aortic valve stenosis (Cardiac disorders) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Leuprorelin Acetate (N=11125)
Injection site erythema (General disorders) | 278
Injection site induration (General disorders) | 904
Hot flush (Vascular disorders) | 247

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be published prior to publication of a multi-center report submitted for publication within 18 months after conclusion or termination of a study at all study sites. Results publications will be submitted to sponsor for review 60 days in advance of publication. Sponsor can require removal of confidential information unrelated to study results. Sponsor can embargo a proposed publication for another 60 days to preserve intellectual property.